CLINICAL TRIAL: NCT04067843
Title: Effects of Photodynamic Therapy on the Human Inguinal Skin Microbiome to Improve Antiseptic Effect - a Pilot Study
Brief Title: Effect of Photodynamic Treatment on Skin Microbiome. Single Center Study
Acronym: PHOMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-005252
Record Dates: First submitted 2019-08-09; First posted 2019-08-28 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Wound Infection Deep Incisional Surgical Site; Prosthesis and Implants; Surgical Site Infection; Prosthetic Joint Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: The investigator will collect scrapings from the skin surface and quantitatively evaluate bacterial species and density before and after photodynamic treatment in combination with skin antisepsis of povidone-iodine/alcohol, in aim 1 immediately after skin antisepsis, and in aim 2, 21 days after photodynamic treatment. For aim 2, the investigators will additionally evaluate changes of sebaceous and sweat glands after photodynamic treatment using histopathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photodynamic treatment (Experimental): Skin microbiome after photodynamic treatment before and after skin antisepsis
  Interventions: Procedure: Photodynamic treatment

INTERVENTIONS:
Procedure: Photodynamic treatment — Photosensitiser application, followed by fluorescence photography Photodynamic therapy (PHT) (1x) over 15 minutes
  Other Names: PDT

SUMMARY:
The overarching aim of this research project is to prevent orthopedic implant-associated infections. This study aims to investigate if photodynamic therapy has an effect on bacterial skin colonization and decrease number of colonizing bacteria associated with sebaceous and sweat glands in order to improve skin antisepsis strategies for the prevention of surgical site infections.

DETAILED DESCRIPTION:
Background. Periprosthetic joint infections are increasing due to our elderly population with the need of a joint prosthesis. These infections are difficult to treat, because bacteria are able to be sessile (biologically inactive) in the biofilms formed within one day on the orthopedic implant surface. Notably, the current available antibiotics do not penetrate the biofilm or are not active against the sessile form of bacteria - rifampicin being the only antibiotic being active. Therefore, prevention is key. In the current paradigm, bacteria from the skin surface or dermis - such as Staphylococcus aureus, coagulase-negative staphylococci, or Cutibacterium sp. - contaminate the peri-implant tissue during surgery. In an ongoing study with the Orthopedic University Hospital Balgrist (manuscript in preparation), the investigators found that the common practice of skin antisepsis is ineffective to eliminate skin bacteria before surgery. Strikingly, the skin bacteria hide in sebaceous or sweat glands. Photodynamic treatment has recently gained attention in the treatment of acne patients, a disease of the pilosebaceous unit, in which also Cutibacterium acnes is implicated. The photodynamic treatment works here on the one hand through a long-lasting destruction of the sebaceous glands, and on the other hand due to anti-inflammatory and antimicrobial effects.

Hypothesis. The investigators hypothesize that photodynamic treatment improves skin antisepsis before surgical implantation of foreign material by reduction of persistent skin colonizing bacteria through the destruction of the sebaceous and sweat glands and by its bactericidal effects Overall and specific objectives. The overarching aim of this research project is to prevent orthopedic implant-associated infections. The specific aim is to evaluate the effect of photodynamic treatment on colonizing bacteria immediately after surgical skin antisepsis (aim 1) and 3 weeks later (aim 2). In aim 3, the investigators will evaluate phylogenetic similarity of same bacterial species before and after photodynamic treatment if they persist.

Methods. The investigators will collect scrapings from the skin surface and quantitatively evaluate bacterial species and density before and after photodynamic treatment in combination with skin antisepsis of povidone-iodine/alcohol, in aim 1 immediately after skin antisepsis, and in aim 2, 21 days after photodynamic treatment. For aim 2, the investigators will additionally evaluate changes of sebaceous and sweat glands after photodynamic treatment using histopathology. To evaluate phylogenetic similarity of same bacterial species before and after photodynamic treatment, the investigators will investigate the core genome using whole genome sequencing.

Relevance and outlook. The current study will investigate if photodynamic treatment is able to improve preoperative skin preparation to decrease surgical site infections in hip arthroplasty surgery. A decrease of implant-associated infections has multiple benefits, among others reduced morbidity, mortality and lower health costs. This study shall provide the fundament for a prospective cohort study of patients with planned hip arthroplasty for investigating the effect of photodynamic treatment before skin antisepsis.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female participants ≥ 18 years who

* volunteer for the pilot study in which a routine photodynamic treatment in the Department of Dermatology will be applied and effect of skin colonization will be analyzed, and
* an informed consent is signed by the participant (after information about the project).

Exclusion Criteria:

* Pregnant and lacting women
* Participants with inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
* Participants taking antibiotics in the 14 days prior to the photodynamic treatment or until follow-up at 21 days
* Participants who received oral retinoid therapy within the last 6 months
* Participants who received anti-inflammatory agents as NSAR within the 14 days prior and after the PDT
* Participants taking any photosensitizing drugs within 4 weeks prior to the photodynamic treatment (PDT)
* Participants who had a history of photosensitivity disorder
* Fitzpatrick's skin phototype V-VI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Achermann, MD, Principal Investigator — University Hospital Zurich, Department of Infectious Diseases and Hospital Epidemiology
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Photodynamic Treatment: Skin microbiome after photodynamic treatment before and after skin antisepsis
  Photodynamic treatment: Photosensitiser application, followed by fluorescence photography, Photodynamic therapy (PDT) (1x) over 15 minutes
- Control Group: Skin microbiome before and after skin antisepsis, no photodynamic treatment
Period: Overall Study
Arm/Group | Photodynamic Treatment | Control Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Photodynamic Treatment: Skin microbiome analysis after photodynamic treatment before and after skin antisepsis
- Control Group: No photodynamic treatment: Skin microbiome before and after skin antisepsis without photodynamic treatment
- Total: Total of all reporting groups
Arm/Group | Photodynamic Treatment | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bacterial Growth Before and After Photodynamic Treatment and After Skin Antisepsis
Description: Skin swabs were taken before photodynamic treatment, after photodynamic treatment and after antisepsis for evaluation of bacterial growth on agar plates
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Photodynamic Treatment: Skin swabs were taken before photodynamic treatment as baseline, after photodynamic treatment and after skin antisepsis to analyse the skin microbiome
  Photodynamic treatment: Photosensitiser application, followed by fluorescence photography, Photodynamic therapy (PDT) (1x) over 15 minutes
- Control Group: Skin swabs were taken before and after skin antisepsis
Arm/Group | Photodynamic Treatment | Control Group
Number analyzed (Participants) | 10 | 10
Participants
  Bacterial growth at baseline | 10 | 10
  Bacterial growth after PDT | 3 | NA — in the control group, skin swabs were only taken before and after antisepsis. PDT was not performed
  Bacterial growth after antisepsis | 0 | 5

2. Primary Outcome: Number of Participants With Bacterial Growth 3 Weeks After Photodynamic Treatment
Description: Skin swabs were taken 21 days after photodynamic treatment before and after skin antisepsis to evaluate bacterial growth on agar plates
Time Frame: Day 21±3 after PDT treatment
Population: was only performed in the photodynamic treatment arm (n=10) and not in the control group
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Treatment
Number analyzed (Participants) | 10
Participants
  Bacterial growth before antisepsis | 10
  Bacterial growth after antisepsis | 6

3. Secondary Outcome: Phylogenetic Comparisons of Isolated Bacteria
Description: was not performed due to clear results in aim 1 and 2.
Time Frame: Day 1 and Day 21
Population: Phylogenetic Comparisons of Isolated Bacteria was not performed due to clear results in aim 1 and 2.
Groups:
- Phylogenetic Comparisons of Isolated Bacteria: was not performed due to clear results in aim 1 and 2.
Arm/Group | Phylogenetic Comparisons of Isolated Bacteria
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from baseline until follow up on day 21
Groups:
- Photodynamic Treatment: Participants were treated with photodynamic treatment
- Control Group: Participants were not treated with photodynamic treatment
Arm/Group | Photodynamic Treatment | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04067843/Prot_SAP_000.pdf